CLINICAL TRIAL: NCT04998903
Title: Role of Fiberoptic Bronchoscopy in Hematopoietic Stem Cell Transplant Patients With Pulmonary Infiltrates in Changing Management Decisions: An Observational Study
Brief Title: Change in Management Following Bronchoscopy in Hematopoietic Stem Cell Transplant Patients With Pulmonary Infiltrates
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr Liju Ahmed, Consultant Pulmonologist, King Faisal Specialist Hospital & Research Center
Other Study IDs: 2141128
Record Dates: First submitted 2021-08-01; First posted 2021-08-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stem Cell Transplant Complications; Pulmonary Complication
Keywords: Stem cell transplant; Hematopoietic Stem Cell; Pulmonary infiltrates; Fiberoptic bronchoscopy
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage (BAL) BAL - cytology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stem cell transplant with Graft versus host disease: Patients who following hematopoietic stem cell transplant suffered from graft versus host disease and presented with pulmonary infiltrates.
  Interventions: Procedure: Fiberoptic Bronchoscopy

INTERVENTIONS:
Procedure: Fiberoptic Bronchoscopy — Fiberoptic bronchoscopy done under conscious sedation
  Other Names: Broncho-alveolar lavage; Transbronchial biopsy

SUMMARY:
Hematopoietic stem cell transplant (HSCT) is a modality that is increasingly utilized to treat various haematological disorders with a varying degree of success. From 2006 to 2019 use of HSCT worldwide has increased from 50,417 to an estimated 1.5 million. Disease relapse, graft versus host disease (GVHD) and infections are the leading causes of morbidity and mortality in patients with HSCT. Pulmonary complications, in particular, are common in patients with HSCT, and the diagnostic approach and management of these complications remain a challenge. FOB is one of the standard and least invasive diagnostic modality for these patients. However, the diagnostic yield and change in clinical decision making in those studies have been variable. Furthermore, all these studies were retrospective, with one exception.

The investigators designed an observational study to understand the rate of change in clinical decision making following Fiberoptic bronchoscopy (FOB). The investigators also looked at the yield of FOB and characteristics associated with a positive diagnostic yield.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplant (HSCT) is a modality that is increasingly utilized to treat various hematological disorders with a varying degree of success. From 2006 to 2019 use of HSCT worldwide has increased from 50,417 to an estimated 1.5 million. Disease relapse, graft versus host disease (GVHD) and infections are the leading causes of morbidity and mortality in patients with HSCT. Pulmonary complications, in particular, are common in patients with HSCT, and the diagnostic approach and management of these complications remain a challenge. Reasons for this possibly include a broad spectrum of etiologies, subtle and insidious clinical manifestations, non-specific radiological features, and limited biomarkers. On the other hand, surgical procedures to obtain lung biopsy, which is the ultimate diagnostic tool, are often contraindicated or present high risks to the patients. In this context, less invasive testing such as fiberoptic bronchoscopy (FOB) deserves further consideration. Previous studies showed that the yield of FOB, a low-risk procedure, may provide helpful information in the post HSCT patient with pulmonary infiltrates. However, the diagnostic yield and change in clinical decision making in those studies have been variable. Furthermore, all these studies were retrospective, with one exception.

The stem cell transplant activity in Saudi Arabia has increased exponentially in recent times, with more than 6000 stem cell transplants performed by 2016. Furthermore, the patient population is different regarding specific genetic and immunologic characteristics, underlying disorders and prevalent opportunistic pathogens. Therefore, this study was designed to prospectively evaluate the diagnostic value of FOB in those patients presenting with pulmonary infiltrates.

Study design and Method

This was a retrospective observational study of all patients who had HSCT and pulmonary infiltrates that required bronchoscopy. Data for demographics, clinical presentation, CT scan characteristics, FOB dates and details, microbiology, virology, cytology, histology, change in clinical decision making before and after FOB and 6 months outcome following bronchoscopy were collected.

Primary outcome

Rate of change in clinical decision making following FOB

Secondary outcome

Clinical characteristics associated with a positive yield in FOB CT scan characteristics associated with a positive yield in FOB Six month outcome of patients following FOB.

Statistics

Descriptive statistics for continuous variables were reported as mean ± standard deviation, and categorical variables were summarized as frequencies and percentages. The median and interquartile range (IQR) was used where appropriate.

Continuous variables were compared by independent Student's t-test/ANOVA or non-parametric (Mann Whitney U/Kruskal Wallis) test as appropriate, while categorical variables were compared by Chi-square test. Fisher's exact probability test was applied when examining variables of low incidence. Logistic regression was used to test the association between dependent and independent variables. The level of significance was set at a p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All patients who suffered from GVHD following Hematopoietic Stem Cell Transplant and had Pulmonary Infiltrate's requiring Fiberoptic Bronchoscopy.

Exclusion Criteria:

* Any patients aged less than 14 years.
* Unable to consent
* Those patients who the primary physician decided not have Fiberoptic Bronchoscopy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was those who had HSCT and suffered from GVHD presenting with pulmonary infiltrates.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Rate of change in clinical decision making following FOB | within 1 months of FOB
  number of patients whose clinical management changed directly as a consequence of fiberoptic bronchoscopy

SECONDARY OUTCOMES:
Clinical characteristics associated with a positive yield in Fiberoptic Bronchoscopy | Within 2 weeks of presentation to FOB
  clinical characteristics associated with a positive microbiology, virology or cytological yield.
CT scan patterns associated with a positive yield in Fiberoptic Bronchoscopy | CT within one month before the FOB
  clinical characteristics associated with a positive microbiology, virology or cytological yield.
Six month outcome of patients following FOB | six months
  Mortality in the six months following FOB.

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Anonymized data of individual participant will be shared.

REFERENCES:
- [Result] Gratwohl A, Pasquini MC, Aljurf M, Atsuta Y, Baldomero H, Foeken L, Gratwohl M, Bouzas LF, Confer D, Frauendorfer K, Gluckman E, Greinix H, Horowitz M, Iida M, Lipton J, Madrigal A, Mohty M, Noel L, Novitzky N, Nunez J, Oudshoorn M, Passweg J, van Rood J, Szer J, Blume K, Appelbaum FR, Kodera Y, Niederwieser D; Worldwide Network for Blood and Marrow Transplantation (WBMT). One million haemopoietic stem-cell transplants: a retrospective observational study. Lancet Haematol. 2015 Mar;2(3):e91-100. doi: 10.1016/S2352-3026(15)00028-9. Epub 2015 Feb 27. PMID 26687803
- [Result] Styczynski J, Tridello G, Koster L, Iacobelli S, van Biezen A, van der Werf S, Mikulska M, Gil L, Cordonnier C, Ljungman P, Averbuch D, Cesaro S, de la Camara R, Baldomero H, Bader P, Basak G, Bonini C, Duarte R, Dufour C, Kuball J, Lankester A, Montoto S, Nagler A, Snowden JA, Kroger N, Mohty M, Gratwohl A; Infectious Diseases Working Party EBMT. Death after hematopoietic stem cell transplantation: changes over calendar year time, infections and associated factors. Bone Marrow Transplant. 2020 Jan;55(1):126-136. doi: 10.1038/s41409-019-0624-z. Epub 2019 Aug 27. PMID 31455899
- [Result] Harris B, Geyer AI. Diagnostic Evaluation of Pulmonary Abnormalities in Patients with Hematologic Malignancies and Hematopoietic Cell Transplantation. Clin Chest Med. 2017 Jun;38(2):317-331. doi: 10.1016/j.ccm.2016.12.008. PMID 28477642
- [Result] Lim DH, Lee J, Lee HG, Park BB, Peck KR, Oh WS, Ji SH, Lee SH, Park JO, Kim K, Kim WS, Jung CW, Park YS, Im YH, Kang WK, Park K. Pulmonary complications after hematopoietic stem cell transplantation. J Korean Med Sci. 2006 Jun;21(3):406-11. doi: 10.3346/jkms.2006.21.3.406. PMID 16778380
- [Result] Lucena CM, Torres A, Rovira M, Marcos MA, de la Bellacasa JP, Sanchez M, Domingo R, Gabarrus A, Mensa J, Agusti C. Pulmonary complications in hematopoietic SCT: a prospective study. Bone Marrow Transplant. 2014 Oct;49(10):1293-9. doi: 10.1038/bmt.2014.151. Epub 2014 Jul 21. PMID 25046219